CLINICAL TRIAL: NCT00182325
Title: Women's Web Access to Their Own Antenatal Health Record and Personalized Health Information: Effect on Pregnancy Health Outcomes and Patient Satisfaction
Brief Title: Effects of a Personalized Web-based Antenatal Care Planner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RDF-160
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Pregnancy
Keywords: medical record; pregnancy; Internet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- personalized web prenatal information (Experimental): Personalized health information for pregnancy through personal health record
  Interventions: Behavioral: personalized web prenatal information
- general web prenatal information (Active Comparator): General pregnancy health related websites
  Interventions: Behavioral: general web prenatal information

INTERVENTIONS:
Behavioral: personalized web prenatal information
  Arms: personalized web prenatal information
Behavioral: general web prenatal information
  Arms: general web prenatal information

SUMMARY:
Many women are turning to the Internet to meet their health information needs, but the large amount of information available, as well as the unknown reliability and applicability of information can be overwhelming. Studies in specific patient populations have determined that patients given access to personalized, on-line medical information are more satisfied with their care than patients provided generalized information. None of these studies have looked at whether this type of patient education would be helpful for pregnant women. This study is being done to determine whether pregnant women who have access to their own health records and personalized health information over the Internet are more satisfied with their prenatal care, and if they are more compliant with health visits and tests, compared to pregnant women who receive only generic pregnancy information on the Internet and from pamphlets

DETAILED DESCRIPTION:
Many women are turning to the Internet to meet their health information needs, but the large amount of information available, as well as the unknown reliability and applicability of information can be overwhelming. Studies in specific patient populations have determined that patients given access to personalized, on-line medical information are more satisfied with their care than patients provided generalized information. None of these studies have looked at whether this type of patient education would be helpful for pregnant women. This study is being done to determine whether pregnant women who have access to their own health records and personalized health information over the Internet are more satisfied with their prenatal care, and if they are more compliant with health visits and tests, compared to pregnant women who receive only generic pregnancy information on the Internet and from pamphlets

Women are being randomly assigned to receive secure access to pregnancy health information links chosen by the centre's physicians, or to receive these links with access to their online personal health that includes the antenatal record and a section of their care planner, from the centre's electronic medical record

ELIGIBILITY:
Inclusion Criteria:

* less than 28 weeks pregnant access to Internet

Exclusion Criteria:

* cannot speak/read English and no translator

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 193 (Actual)
Dates: Start 2004-02 (Actual); Primary Completion 2006-08 (Actual); Study Completion 2006-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather Waters, MD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Personalized Information and Internet Access: Women in this group were given access to their own personal antenatal health record and personalized information through the clinic's antenatal care planner, as well as access to the study site website, which provided links to pregnancy information that was pre-approved by the study team.
- General Resource Internet Access: Women in this group were given access to the study site website, which provided links to pregnancy information that was pre-approved by the study team
Period: Overall Study
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
Started | 97 | 96
Completed | 63 (63 completed survey, 85 included in intention-to-treat analysis) | 43 (43 completed survey, 89 included in intention-to-treat analysis)
Not Completed | 34 | 53
Not completed — Lost to Follow-up | 7 | 7
Not completed — Miscarriage | 5 | 3
Not completed — Did not complete survey | 22 | 43

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access | Total
Number analyzed (Participants) | 97 | 96 | 193
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.7 (5.3) | 26.4 (5.6) | 27.1 (5.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 96 | 193
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Married or common-law [Count of Participants; unit: Participants] — Population: Full demographic information was available only for the women who completed the surveys.
  Participants
    number analyzed (Participants) | 95 | 92 | 187
    (all) | 75 | 72 | 147
Primiparous [Count of Participants; unit: Participants] — Population: Full demographic information was available only for the women who completed the surveys.
  Participants
    number analyzed (Participants) | 93 | 93 | 186
    (all) | 60 | 64 | 124
At least some post-secondary education [Count of Participants; unit: Participants] — Population: Full demographic information was available only for the women who completed the surveys.
  Participants
    number analyzed (Participants) | 91 | 90 | 181
    (all) | 58 | 59 | 117

OUTCOME MEASURES:

1. Primary Outcome: Uptake of Service
Description: Number of log-ins
Time Frame: 11 months
Population: An intention-to-treat analysis was conducted. Participants were included in the analysis that started or completed the survey and excludes participants that were lost to follow-up or had a miscarriage.Intervention group: 63 completed survey + 22 partially complete survey =85). Control group: 53 completed survey + 43 partially complete survey = 96).
Measure: Mean (Standard Deviation); unit: Log-ins
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
Number analyzed (Participants) | 85 | 89
Log-ins | 10.4 (17.8) | 1.8 (1.4)
Statistical Analysis 1: Comparison: Personalized Information and Internet Access vs General Resource Internet Access; Test type: Superiority; p < 0.0001, t-test, 2 sided

2. Primary Outcome: Easy to Log on
Description: Women were asked to rate their agreement with statements about the website from strongly agree (1) to strongly disagree (5) on a five-point scale. Results presented here are mean responses to questionnaire about the pregnancy website in the two randomized groups.
Time Frame: 11 months
Population: The number of completed surveys was 63 (64.9%) in the personalized information and Internet access group, and 43 (44.8%) in the general resource Internet access group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
Number analyzed (Participants) | 63 | 43
score on a scale | 1.4 (0.5) | 1.5 (0.9)
Statistical Analysis 1: Comparison: Personalized Information and Internet Access vs General Resource Internet Access; Test type: Superiority; p = 0.84, t-test, 2 sided

3. Primary Outcome: Information Easy to Understand
Description: as for outcome 2
Time Frame: 11 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
Number analyzed (Participants) | 63 | 43
score on a scale | 1.4 (0.5) | 1.5 (0.6)
Statistical Analysis 1: Comparison: Personalized Information and Internet Access vs General Resource Internet Access; Test type: Superiority; p = 0.68, t-test, 2 sided

4. Primary Outcome: Learned Something New
Description: as for outcome 2
Time Frame: 11 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
Number analyzed (Participants) | 63 | 43
score on a scale | 1.8 (0.9) | 1.9 (0.8)
Statistical Analysis 1: Comparison: Personalized Information and Internet Access vs General Resource Internet Access; Test type: Superiority; p = 0.67, t-test, 2 sided

5. Primary Outcome: Easy to Find Information
Description: as for outcome 2
Time Frame: 11 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
Number analyzed (Participants) | 63 | 43
score on a scale | 1.9 (0.9) | 1.8 (0.7)
Statistical Analysis 1: Comparison: Personalized Information and Internet Access vs General Resource Internet Access; Test type: Superiority; p = 0.57, t-test, 2 sided

6. Primary Outcome: Helped me Stay Healthy
Description: as for outcome 2
Time Frame: 11 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
Number analyzed (Participants) | 63 | 43
score on a scale | 1.8 (0.8) | 1.6 (0.7)
Statistical Analysis 1: Comparison: Personalized Information and Internet Access vs General Resource Internet Access; Test type: Superiority; p = 0.17, t-test, 2 sided

7. Primary Outcome: Helped me Learn About Risks
Description: as for outcome 2
Time Frame: 11 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
Number analyzed (Participants) | 63 | 43
score on a scale | 1.9 (0.8) | 1.8 (0.8)
Statistical Analysis 1: Comparison: Personalized Information and Internet Access vs General Resource Internet Access; Test type: Superiority; p = 0.46, t-test, 2 sided

8. Primary Outcome: Helped me Understand Tests
Description: as for outcome 2
Time Frame: 11 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
Number analyzed (Participants) | 63 | 43
score on a scale | 1.7 (0.7) | 1.6 (0.8)
Statistical Analysis 1: Comparison: Personalized Information and Internet Access vs General Resource Internet Access; Test type: Superiority; p = 0.57, t-test, 2 sided

9. Primary Outcome: Helped me Make Decisions
Description: as for outcome 2
Time Frame: 11 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
Number analyzed (Participants) | 63 | 43
score on a scale | 2.1 (0.9) | 2.4 (1.2)
Statistical Analysis 1: Comparison: Personalized Information and Internet Access vs General Resource Internet Access; Test type: Superiority; p = 0.26, t-test, 2 sided

10. Primary Outcome: Helped me Remember Appointments
Description: as for outcome 2
Time Frame: 11 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
Number analyzed (Participants) | 63 | 43
score on a scale | 2.9 (1.3) | 3.5 (1.4)
Statistical Analysis 1: Comparison: Personalized Information and Internet Access vs General Resource Internet Access; Test type: Superiority; p = 0.12, t-test, 2 sided

ADVERSE EVENTS:
Arm/Group | Personalized Information and Internet Access | General Resource Internet Access
All-Cause Mortality (participants affected / at risk) | 0/97 | 0/96
Serious Adverse Events (participants affected / at risk) | 0/97 | 0/96
Other Adverse Events (participants affected / at risk) | 0/97 | 0/96

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No